CLINICAL TRIAL: NCT00094562
Title: AAFA™ Fish Oil Nutritional Supplementation to Maintain Body Weight in Patients With Disease-Related Weight Loss
Brief Title: A Fish Oil Supplement to Maintain Body Weight in Patients With Disease-Related Weight Loss
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: J0275; 03-02-10-12 (Other: JHM IRB); P50AT000437 (NIH)
Record Dates: First submitted 2004-10-20; First posted 2004-10-21 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2008-04

CONDITIONS: Cancer; Cancer Cachexia; Chronic Obstructive Pulmonary Disease; Chronic Heart Failure; Rheumatoid Arthritis
Keywords: Cancer; Cancer Cachexia; Weight Loss; Chronic Obstructive Pulmonary Disease; Chronic Heart Failure; Rheumatoid Arthritis
MeSH Terms: conditions — Neoplasms; Pulmonary Disease, Chronic Obstructive; Arthritis, Rheumatoid; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Fish oil supplement

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of fish oil supplements in maintaining weight in people with disease-related weight loss and/or cachexia.

DETAILED DESCRIPTION:
The overall goal of this project is to evaluate the safety and efficacy of nutritional supplementation with fish oils to maintain weight in patients with disease-related weight loss (cachexia). Weight loss commonly results in a poorer prognosis, functional status, and quality of life. Despite the high morbidity and mortality associated with cachexia, mainstream treatment does not sustain weight and although nutritional supplements are commonly used, many of these have not been tested in clinical trials. Recent work in cachexia has revealed that this is mediated by pro-inflammatory cytokines. There are data that suggests that fish oils can affect the underlying pathogenic inflammatory response and have an affect on weight maintenance and nutritional balance

Diseases in which cachexia is most common:

* Cancer
* Chronic Heart Failure (CHF)
* Chronic Obstructive Pulmonary Disease (COPD)
* Rheumatoid Arthritis (RA)

Goals of the Study:

* To evaluate the safety and efficacy of fish oils vs. corn oil in the maintenance of weight and lean body mass in patients with disease-related weight loss.
* To understand the mechanism of fish oil effect on health maintenance by evaluating the anti-inflammatory, anti-catabolic, anti-oxidant and anabolic actions of these compounds
* To document the effect of our interventions on quality of life and functional status.

Study Outline:

Participants will be randomly assigned to receive either fish oil supplements or corn oil for the duration of this 3-month study. Participants will have five study visits and two telephone interviews. During each study visit, participants will undergo laboratory tests, a physical exam, and a dual energy X-ray absorptiometry (DEXA) bone scan. Participants will be asked to keep a food diary during the study. During the telephone interviews, participants will be asked health-related questions and discuss their current functional status.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women with disease-related weight loss e.g. cardiac cachexia, COPD, CHF, RA.
* All stages of Pancreatic cancer patients (No weight loss requirements)
* All stages of cancer with 5% weight loss
* At least 6 weeks post-surgery
* On a stable dose of medications for at least 6 weeks prior to study entry
* Most recent ECOG Performance status score of 0,1,2,or 3 if applicable
* Agree to use acceptable methods of contraception during the study and for 3 months after study completion, for female participants. Females with reproductive potential must have a negative urine or serum pregnancy test within 7 days of study.
* Willing to continue current therapy for cancer for the duration of the study
* If with diabetes mellitus HgbA1C of <10%
* Adequate bone marrow function ANC> 1000/mm3, platelets 50,000/mm3, hemoglobin, 8g/dl.
* No active infections including known history of HIV or viral hepatitis.

Exclusion Criteria:

* Esophageal Cancer
* Individuals with hypertriglyceridemia
* Life expectancy of less than 12 weeks
* Alcohol consumption more than 3 drinks/day for men or 2 drinks/day for women.
* Untreated endocrine problems
* Severe Depression
* Untreated endocrine problems, such as hypothyroidism. Gonadal dysfunction from a known primary endocrine dysfunction (e.g. Klinefelters syndrome, pituitary tumor, testicular neoplasms, testicular surgery.
* Medications that impair sex hormone synthesis, secretion, or function (e.g. spironolactone, anti-estrogens, anabolic steroids and androgens.
* Fish oils within 3 months prior to study entry.
* Any infectious disease, such as HIV or viral hepatitis.
* Vitamins in doses greater than the Recommended Daily Allowance (RDA)
* Herbs in the month prior to study entry.
* Only participation in other cachexia studies is prohibited.
* Prothrombin Time INR > 2.5 on Coumadin and INR > 2.0 not on Coumadin.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2004-06; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Body weight
lean body mass

CONTACTS AND LOCATIONS:
Overall Officials: Adrian S. Dobs, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States